CLINICAL TRIAL: NCT01582464
Title: Effect of Social Marketing on Attitudes Towards Protective Headwear in Older Adults to Reduce Traumatic Brain Injury
Brief Title: Addressing Attitudes to Improve Use of Protective Headwear in Older Adults
Acronym: AAIU-PHOA
Status: Completed | Type: Observational
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Steven C. Castle, MD, Principle Investigator, University of California, Los Angeles
Other Study IDs: 2010-012
Record Dates: First submitted 2012-04-18; First posted 2012-04-20 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Injury of Unknown Intent Due to Fall From Height; Traumatic Brain Injury
Keywords: Protective Headwear; Social Marketing; Theory of Planned Behavior
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Social Marketing; Head Protective Devices

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Older Adults in a Senior Community: Residents of a Continuing Care Retirement Community (CCRC) that is a part of The Be Group (previously known as Southern California Presbyterian Homes), with no exclusion other than being able to communicate in English and provide consent to participate.
  Interventions: Behavioral: Social Marketing for protective headgear

INTERVENTIONS:
Behavioral: Social Marketing for protective headgear — Social marketing was done using a CQI manner after each focus group with experts and with seniors using a structured interview approach with an iterative process to develop a progressive method of presenting information about head injuries and their input on a new prevention.
  To measure changes in attitudes, the participants were given an attitudes questionnaire (PHAQ), & a demographic & functional status questionnaire. Input into the social marketing content was sought in a structured interview manner, and by using an audience response system with questions projected by power point. At the conclusion of the social marketing, the PHAQ was repeated and sent to participants 2 weeks after the focus group to gage stability of changes in attitudes.
  Other Names: SMARTY and commercially available protective Headgear

SUMMARY:
The goal of this phase of the project is to identify the elements of the Theory of Planned Behavior (TPB) that should be targeted to provide the most influence on older adults' behavior (or other stakeholders) to purchase and wear protective headwear. The investigators also intend to determine the format of communication (social marketing/academic detailing) that is most influential for different key stakeholder groups. The TPB has been useful in understanding behavior change related to exercise and adaptive equipment use (such as grab bars, canes, hip protectors); in understanding how a person's attitudes, subjective/social norms and perceived behavioral control inform the development of intention that leads to behavior change.

DETAILED DESCRIPTION:
1. Design of Social Marketing/Consumer Preferences Trial

   a. Development of Protective Headwear Attitudes Questionnaire To develop a questionnaire specific to attitudes about protective headwear, the authors reviewed existing papers that applied the Theory of Planned Behavior to other health behaviors such as the use of canes or walkers and adherence to exercise. Questions were drafted to address attitudes (24), subjective norms (14) and perceived behavioral control (14) about the behavior of using protective headwear. The rationale and specific questions were presented to an expert panel and clinicians (behavioralist, 3 geriatricians, long-term care nurse and a nurse health services researcher) to evaluate the content and face validity of each question, and to rank each as high or low importance within each domain. Item reduction and refinement following the expert panels identified 26 candidate questions. Analysis of the PHAQ as an instrumented was also completed
2. Social Marketing Approach

   1. Expert panel Input on social marketing materials Input on the social marketing phase was conducted on two focus groups of 6 clinicians, geriatricians and nurses, and the social marketing tools were updated and improved in a CQI manner after each focus group with experts and with seniors in retirement communities. Please review transcripts on the input from seniors.
   2. Social Marketing Focus groups/Process The social marketing approach was developed and refined using a structured interview approach with each focus group of older adults. A total 6 focus groups were conducted at 4 communities with a total of 36 participants. An iterative process was used to improve the content of the social marketing after each session.

      The goal was to develop a progressive method of presenting information about the magnitude of head injuries and the development of a new product that we wanted their input towards the final design. The progression was done with First, a one page flier, Second, a three minute video tape and Finally, a two page article that was patterned after articles that appear in AARP magazine. The flier provided basic information about the risk of TBI and the development of a new product called SMARTY®, which is made of advanced materials so that it is lightweight and can be styled to match the needs of the user and setting. The Video included the discussion of the unrecognized public health issue by one of the authors (SC), photos of the advanced materials and how they work to provide protection, a videotape of the testing of the protective headwear by dropping a crash test dummy and finally the testimonial of the user of a prototype by a colleague who has a seizure disorder. The paper provides more detail and includes a graph of the rapid increase in deaths from TBI in older adults 75 years and over, and a drawing that describes the characteristics of the advanced materials.
   3. Ability to change attitudes To measure changes in attitudes, the participants were given the PHAQ, as well as the demographic and functional status questionnaire when they arrived for the focus group. Input into the social marketing content was sought in a structured interview manner, and by using an audience response system with questions projected by power point. At the conclusion of the social marketing, the PHAQ was repeated and sent to participants 2 weeks after the focus group to gage stability of changes in attitudes.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* >= 65 years old
* Male or Female
* Competent to give informed consent

Exclusion Criteria:

* Non-English Speaking
* Not competent to give informed consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: The population is English speaking male or female > 65 years of age who are competent to give informed consent.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-05; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Castle, MD, Principal Investigator — University of California, Los Angeles
Locations (1):
- Be.Group Facilities, Multiple, California, United States

IPD SHARING:
Plan to Share IPD: No
all data shared will be de-identified